CLINICAL TRIAL: NCT02494102
Title: A Randomized, Double Blind, Placebo Controlled Evaluation of Modafinil vs Placebo for the Treatment of General Anesthesia Related Delayed Emergence in Patients With the Diagnosis of Obstructive Sleep Apnea
Brief Title: Evaluation of Modafinil vs Placebo for Treatment of Anesthesia Delayed Emergence in Obstructive Sleep Apnea
Acronym: ModOSA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Zyad J. Carr, M.D., Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPITALSTUDY00002957
Record Dates: First submitted 2015-07-01; First posted 2015-07-10 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Obstructive Sleep Apnea; Delayed Emergence From Anesthesia
Keywords: Obstructive Sleep Apnea; General Anesthesia; Modafinil
MeSH Terms: conditions — Sleep Apnea, Obstructive; Delayed Emergence from Anesthesia | interventions — Modafinil

STUDY DESIGN:
Intervention Model Description: double blind randomized placebo controlled trial
Who Masked: Participant, Investigator
Masking Description: Computer generated randomization list, subject, clinical team and research team blinded to intervention
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Administered Placebo day of surgery immediately prior to general anesthesia and surgery
  Interventions: Drug: Placebo
- Intervention (Active Comparator): Administered Modafinil 200mg day of surgery prior to general anesthesia and surgery
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — Atypical Psychomotor stimulant
  Other Names: Armodafinil; Provigil
  Arms: Intervention
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether modafinil use in patients with obstructive sleep apnea will improve postoperative delayed emergence after general anesthesia.

DETAILED DESCRIPTION:
This is a randomized, double blind placebo controlled evaluation of modafinil versus placebo for the treatment of general anesthesia related delayed emergence in patients with the diagnosis of obstructive sleep apnea. 124 patients will be recruited and randomized on the day of surgery to receive 200mg modafinil or placebo. After randomization, patients will proceed to the operative suite for surgical procedure under general anesthesia. The primary outcome measured will be post-anesthesia care unit length of stay. Secondary outcomes will include performance on a post-anesthesia recovery scale.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Meets diagnostic criteria for obstructive sleep apnea
3. Willing and able to comply with study procedures
4. Willing and able to provide informed consent
5. If female, not pregnant or lactating and willing to use an acceptable method of barrier birth control (e.g. condoms) for one month after surgery and discontinuation of study medication (modafinil may reduce the effectiveness of steroidal contraception for one month after discontinuation)

Exclusion Criteria:

1. Have a medical condition that, in the study physician's judgment, may interfere with safe participation (active cardiac conditions such as angina, recent myocardial infarction w/in 6 months, severe renal or liver disease, unstable diabetes, or elevated liver enzymes greater than twice normal).
2. Have a current neurological disorder (e.g. organic brain disease, dementia) or major psychiatric condition that would impair the collection of data (schizophrenia, bipolar illness).
3. Currently on prescription medication that is known to interact with the study drug. (ethinylestradiol and triazolam).
4. Have current dependence on cocaine, methamphetamine, alcohol or benzodiazepines (DSM-IV criteria).
5. Have a history of severe valvular heart disease, severe left ventricular hypertrophy, cardiac arrhythmias, angina, cardiac syncope, or pre-syncope or myocardial infarction <6 months.
6. Have a history of uncontrolled or poorly controlled essential hypertension, or a heart rate greater than 70% of the maximum heart rate expected for their age (Formula: 0.70(220 - age).
7. Any condition, in the opinion of the principal investigators that would compromise patient safety.
8. A documented history of sensitivity to modafinil.
9. Current Modafinil use for daytime somnolence associated with obstructive sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zyad J Carr, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Minzenberg MJ, Carter CS. Modafinil: a review of neurochemical actions and effects on cognition. Neuropsychopharmacology. 2008 Jun;33(7):1477-502. doi: 10.1038/sj.npp.1301534. Epub 2007 Aug 22. PMID 17712350
- [Background] Moldofsky H, Broughton RJ, Hill JD. A randomized trial of the long-term, continued efficacy and safety of modafinil in narcolepsy. Sleep Med. 2000 Apr 1;1(2):109-116. doi: 10.1016/s1389-9457(99)00014-3. PMID 10767651
- [Background] Jasinski DR, Kovacevic-Ristanovic R. Evaluation of the abuse liability of modafinil and other drugs for excessive daytime sleepiness associated with narcolepsy. Clin Neuropharmacol. 2000 May-Jun;23(3):149-56. doi: 10.1097/00002826-200005000-00004. PMID 10895398
- [Background] Jasinski DR. An evaluation of the abuse potential of modafinil using methylphenidate as a reference. J Psychopharmacol. 2000 Mar;14(1):53-60. doi: 10.1177/026988110001400107. PMID 10757254
- [Background] Wisor JP, Nishino S, Sora I, Uhl GH, Mignot E, Edgar DM. Dopaminergic role in stimulant-induced wakefulness. J Neurosci. 2001 Mar 1;21(5):1787-94. doi: 10.1523/JNEUROSCI.21-05-01787.2001. PMID 11222668
- [Background] Arnulf I, Homeyer P, Garma L, Whitelaw WA, Derenne JP. Modafinil in obstructive sleep apnea-hypopnea syndrome: a pilot study in 6 patients. Respiration. 1997;64(2):159-61. doi: 10.1159/000196661. PMID 9097352
- [Background] Pack AI, Black JE, Schwartz JR, Matheson JK. Modafinil as adjunct therapy for daytime sleepiness in obstructive sleep apnea. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1675-81. doi: 10.1164/ajrccm.164.9.2103032. PMID 11719309
- [Background] Larijani GE, Goldberg ME, Hojat M, Khaleghi B, Dunn JB, Marr AT. Modafinil improves recovery after general anesthesia. Anesth Analg. 2004 Apr;98(4):976-981. doi: 10.1213/01.ANE.0000108485.29288.B4. PMID 15041583
- [Background] Galvin E, Boesjes H, Hol J, Ubben JF, Klein J, Verbrugge SJ. Modafinil reduces patient-reported tiredness after sedation/analgesia but does not improve patient psychomotor skills. Acta Anaesthesiol Scand. 2010 Feb;54(2):154-61. doi: 10.1111/j.1399-6576.2009.02093.x. Epub 2009 Aug 31. PMID 19719817

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 patients violated the study protocol and were excluded from the study. Exclusions included Day of Surgery refusal of study medication, surgical case cancellation, and surgeon refusal to participate.
Groups:
- Placebo: Administered Placebo day of surgery immediately prior to general anesthesia and surgery
  Placebo
- Modafinil: Administered Modafinil 200mg day of surgery prior to general anesthesia and surgery
  Modafinil: Atypical Psychomotor stimulant
Period: Overall Study
Arm/Group | Placebo | Modafinil
Started | 42 | 47
Completed | 42 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 patients violated the study protocol and were excluded from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Modafinil | Total
Number analyzed (Participants) | 42 | 47 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (13) | 54 (13) | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 23 | 23 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Surgery Type [Count of Participants; unit: Participants] — Proportions by surgical procedure: abdominal surgery, orthopedic surgery, gynecology, otolaryngology, ophthalmology.
  Participants
    abdominal surgey | 27 | 30 | 57
    orthopedic surgery | 2 | 5 | 7
    gynecology | 4 | 7 | 11
    otolaryngology | 8 | 5 | 13
    opthalmology | 1 | 0 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight in kilograms divided by the square of height in meters. This variable was measured preoperatively prior to intervention.
  kg/m^2 | 38.2 (11.1) | 44.9 (11.6) | 41.9 (11.3)
Hypertension [Number; unit: participants] — number of participants with the diagnosis of hypertension
  participants | 26 | 33 | 59
History of Delayed Emergence [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Length of Time From Extubation to Discharge From Postanesthesia Recovery Unit
Description: Length of time of above compared between groups
Time Frame: 24 hours
Population: 16 participants violated the study protocol
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Placebo | Modafinil
Number analyzed (Participants) | 42 | 47
minutes | 53.5 [41 to 80] | 61.0 [46 to 91]

2. Secondary Outcome: Postanesthesia Quality Recovery Scale Score
Description: Postanesthesia quality recovery scale (PQRS). Component and aggregate scoring on the scale. Measures physiology, nociceptive, emotional activities of daily living cognitive and overall patient perspective. The scale is dimensionless and the aggregate of all individually tested dimensions is scaled from 17-65. A higher value implies improved postanesthesia recovery. Mean difference was assessed in each patient and aggregated thus patients with no difference between pre- and post-operative scores were zeroed (received a zero score if the difference was zero). A negative value was associated with worse outcome.
Time Frame: baseline and 6 hours after surgery
Population: 16 patients violated study protocol and were excluded
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Modafinil
Number analyzed (Participants) | 42 | 47
units on a scale | -5.67 (4.74) | -8.91 (7.98)

ADVERSE EVENTS:
Time Frame: Perioperative time period (within 24 hours)
Arm/Group | Placebo | Intervention
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/47
Other Adverse Events (participants affected / at risk) | 0/42 | 0/47

LIMITATIONS AND CAVEATS:
Trial terminated for statistical futility on scheduled interim analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT02494102/Prot_SAP_000.pdf